CLINICAL TRIAL: NCT03370809
Title: Assessment of Positron Emission Tomography to Early Detect Frailty in Onco-geriatry
Acronym: FOGTEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Antoine VERGER, MD, PhD, Central Hospital, Nancy, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PSS2017/FOGTEP-VERGER/VS
Record Dates: First submitted 2017-12-07; First posted 2017-12-12 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Patients Over 75 Years Old With a Cancer Discovery
Keywords: Frailty; Oncogeriatric; PET 18F-FDG; SPM (Statistical Parametric Mapping); Neurology
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients over 75 years old with cancer discovery (Experimental): Elderly patients with cancer have a 18F-FDG PET whole body performed routinely in the initial assessment . A cerebral recording is added 45 minutes after the 18F-FDG injection and just before the registered whole body
  Interventions: Radiation: Brain PET/CT step

INTERVENTIONS:
Radiation: Brain PET/CT step — a cerebral PET/CT will be registered on the 45th minute after 18F-FDG injection and just before the whole body recording. This recording does'nt need a new injection but needs a low dose scanner

SUMMARY:
Oncogeriatric frailty assessment is a multifactorial approach to determine the most appropriate treatment for the health status of elderly cancer patients and this assessment is recommended for patients over 75 years of age.

Oncogeriatric frailty is based on the SIOG-2 (International Society of Geriatric Oncology-2) clinical scale (assessing comorbidities, autonomy, nutrition, cognitive and thymic domains) defining 3 levels of frailty: (1) harmonious aging, (2) vulnerability (reversible stage), (3) fragility (irreversible stage).

So,the management of very old or very frailty patients with poor tolerance or compliance to treatment, often requires to defer standard treatment and monitoring procedures. That is detrimental to these patients prognosis. By contrast with elderly or very old patients without frailty criteria, could benefit from more efficient procedures.

More generally, frailty is associated directly with a cerebral impact on a cognitive or thymic status or indirectly with the cognitive or thymic impacts related with other components (nutritional or autonomy or walking poor status, comorbidities) 18F-Fluorodeoxyglucose (18F-FDG) Positron Emission Tomography (PET), is routinely performed in follow-up cancer patients in most cases, including older patients, to detect neoplastic localizations on the whole body. It also accurately quantifies cerebral glycolytic metabolism when early brain recording is performed. Brain metabolism reflects the neuronal synaptic activity. It is generally decreased in particular brain areas due of neurodegenerative damage with a little or no symptom, of thymic involvement particular in depression or during accelerated cerebral aging of vascular origin. The impairment of the brain function of the elderly, as evidenced by 18F-FDG PET, is most often multifactorial, as frailty. Above all, brain changes are visualized with 18F-FDG PET much earlier than using neuropsychological tests, especially for cognitive impairment.

Our hypothesis is that with 18F-FDG PET, performed routinely in the initial assessment in elderly patients with cancer, it is also possible to obtain reliable and objective parameters of brain function and frailty. 18F-FDG PET is already used to identify cognitive and thymic impairment. This exam would help to assess the frailty and to adapt as best oncologic treatments some of which can also be neurotoxic. 18F-FDG PET is therefore related to brain function in frail patients

ELIGIBILITY:
Inclusion Criteria:

* patients who are more than 75 years old with written informed consent
* patients referred for 18F-FDG PET in an oncological disease newly diagnosed
* patients insured under social security

Exclusion Criteria:

* patients with disease in final stage and life expectancy less than 6 months
* patients under guardianship or curators
* patients with abnormal neurological tests: MMS< 27, with neoplastic or other brain lesions or showing ischemic or cerebral stroke damage
* confused or agitated patient unable to realize a PET
* radiotherapy ou chemiotherapy one year at least of the patient enrollment

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 37 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2022-05-24 (Actual); Study Completion 2022-08-10 (Actual)

PRIMARY OUTCOMES:
Volume of brain with damages detected by quantitative analysis SPM (Statistical Parametric Mapping) | through the completion of the study on average 24 months
  Metabolism of PET cerebral images and correlation with different groups of frailty at the initial visit

SECONDARY OUTCOMES:
Volume of brain with damages detected by quantitative analysis SPM between 2 patient's group with MMSE (MiniMental State Examination) results and threshold value as 24 | 20 months, according to the results of neurology tests at the initial visit and at the 6 month
  Metabolism of PET cerebral images and correlation into 2 frailty groups defined by their results MMSE (MiniMental State Examination) test : group 1 with MMSE < or = 24 and group 2 with MMSE>24, at the initial visit and at the 6 month visit
Volume of brain with damages detected by quantitative analysis SPM between 2 patient's groups with GDS (Geriatric Depression Scale) results and threshold value as 5 | 20 months, according to the results of neurology tests at the initial visit and at the 6 month
  Metabolism of PET cerebral images and correlation into 2 frailty groups defined by their results GDS (Geriatric Depression Scale) test : group 1 with GDS < or = 5 and group 2 with GDS>5 at the initial visit and at the 6 month visit
Volume of brain with damages detected by quantitative analysis SPM between different groups according to the SIOG-2 scale | 20 months, according to the results of neurology tests at the initial visit and at the 6 month
  Metabolism of PET cerebral images and correlation into different patients groups according to the SIOG-2 scale during the geriatric visit over 6 months
Volume of brain with damages detected by quantitative analysis SPM between 2 patient's groups according to an unscheduled hospitalisation over 6 months or no | 20 months,according to the results of neurology tests at the initial visit and at the 6 month
  Metabolism of PET cerebral images and correlation into 2 patients groups with known frailty or no defined by an unscheduled hospitalisations at 6 months
Volume of brain with damages detected by quantitative analysis SPM between 2 patient's groups according to non cancer related death at 12 months or no | 24 months,according to the death or not of the patients asked 12 months after the inclusion
  Metabolism of PET cerebral images and correlation with known excess frailty or no defined by a death non cancer related at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Antoine VERGER, MD, PhD, Principal Investigator — CHRU NANCY, IADI INSERM U1254
Locations (1):
- CHRU NANCY Brabois, nuclear medicine department, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: Undecided